CLINICAL TRIAL: NCT01355302
Title: An Open-Label, Multicenter, Randomized, Phase Ib/II Study of E7050 in Combination With Cisplatin and Capecitabine Versus Cisplatin and Capecitabine Alone in Patients With Advanced or Metastatic Solid Tumors and Previously Untreated Gastric Cancer
Brief Title: E7050 in Combination With Cisplatin and Capecitabine Versus Cisplatin and Capecitabine Alone in Patients With Advanced or Metastatic Solid Tumors and Previously Untreated Gastric Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sites not recruiting
Sponsor: Eisai Inc. (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7050-703; 2011-000774-58 (EudraCT Number)
Record Dates: First submitted 2011-05-16; First posted 2011-05-18 (Estimated); Results first posted 2017-03-13 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-03

CONDITIONS: Advanced or Metastatic Solid Tumors; Previously Untreated Gastric Cancer
Keywords: Cancer; Solid Tumors; Gastric; Phase I; Phase II
MeSH Terms: conditions — Neoplasms | interventions — N-(2-fluoro-4-((2-(4-(4-methylpiperazin-1-yl)piperidin-1-yl)carbonylaminopyridin-4-yl)oxy)phenyl)-N'-(4-fluorophenyl)cyclopropane-1,1-dicarboxamide; Cisplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase Ib: Cohort 1 and 2 and 3 (Experimental): Phase Ib: Cohort 1; 200 mg E7050 + 80 mg/m2 cisplatin + 1000 mg/m2 capecitabine
  Cohort 2; 300 mg E7050 + 80 mg/m2 cisplatin + 2000 mg/m2 capecitabine Cohort 3; 400 mg E7050 + 80 mg/m2 cisplatin + 2000 mg/m2 capecitabine
  Interventions: Drug: E7050; Drug: cisplatin; Drug: capecitabine
- Phase II: Arm 1; E7050 + cisplatin+ capecitabine (Active Comparator): Phase II: Arm 1; MTD E7050 + 80 mg/m2 cisplatin + 2000 mg/m2 capecitabine
  Interventions: Drug: E7050; Drug: cisplatin; Drug: capecitabine

INTERVENTIONS:
Drug: E7050 — E7050 given orally at either 200, 300, or 400 mg once daily.
Drug: cisplatin — Cisplatin will be administered at 80 mg/m2 by intravenous infusion over 60 minutes on Day 1 of each 21-day treatment cycle.
Drug: capecitabine — Capecitabine will be administered at 1000 mg/m2 orally, twice daily (2000 mg/m2 total daily dose) on Days 1 through 14 of each 21-day treatment cycle.

SUMMARY:
The purpose of this study is to determine the following: 1. Find the maximum tolerated dose of E7050 when given in combination with cisplatin and capecitabine in patients with advance or metastatic solid tumors, and 2) Whether E7050 in combination with cisplatin and capecitabine is more effective in patients with previously untreated gastric cancer versus cisplatin and capecitabine alone.

DETAILED DESCRIPTION:
This open-label, multicenter, randomized study will consist of 2 phases:

Phase Ib: a safety run-in period with 3 ascending doses of E7050 in combination with fixed doses of Cisplatin and Capecitabine. This phase will enroll approximately 10 to 15 patients.

* Phase II: a randomized 2-arm design which will enroll 80 patients.

In the phase II portion, Patients will receive study treatment , E7050 in combination with Cisplatin and Capecitabine versus Cisplatin and Capecitabine Alone) for approximately six 21-day cycles (18 weeks). Beyond 18 weeks, patients who are experiencing clinical benefit may continue E7050, with or without Capecitabine (Arm 1), or may continue Capecitabine alone (Arm 2), depending on the original randomization treatment arm. Patients will continue treatment for as long as clinical benefit is sustained and the treatment is well tolerated, until the occurrence of progressive disease (PD), unacceptable toxicity, withdrawal of consent, or withdrawal by investigator, whichever occurs first. Patients will participate in either phase Ib or phase II.

ELIGIBILITY:
Inclusion Criteria

* Histologically confirmed, unresectable, locally advanced or metastatic gastric cancer, including adenocarcinoma of the gastroesophageal junction (Phase II). For the Phase Ib portion, any unresectable, locally advanced or metastatic solid tumor;
* ECOG PS of 0-1;
* Blood pressure must be well-controlled. Patients must have no history of hypertensive crisis or hypertensive encephalopathy; Adequate end organ function

Exclusion Criteria

* Gastric cancer patients who have had a complete gastrectomy;
* Patients with known HER2 over-expressing advanced or metastatic gastric cancer;
* Previously received E7050, its chemical derivatives, anti-cMet, anti-angiogenic therapy, (prior anti-angiogenic therapy is permitted in Phase Ib only).
* For Phase Ib prior systemic therapy is allowed as long as PS and end organ function meet entry criteria;
* For Phase II no prior palliative chemotherapy is permitted. Adjuvant/neoadjuvant chemotherapy is permitted if less than 12 months have elapsed between the end of adjuvant/neoadjuvant therapy and first recurrence;
* Known central nervous system lesions, except for asymptomatic non-progressing, treated brain metastases. Treatment for brain mets, but have been completed at least 4 weeks prior to Day 1
* Palliative radiotherapy is not permitted throughout the study period. Prior palliative radiotherapy within 30 days prior to commencing study treatment;
* Clinically significant hemoptysis;
* Patients with known dihydropyrimidine dehydrogenase deficiency;
* Patients with clinically significant hearing loss that may be further diminished by treatment with cisplatin plus capecitabine (significance of hearing loss to be determined by the Investigator;
* Serious non-healing wound, ulcer, or active bone fracture;
* Major surgical procedure, open biopsy, or significant traumatic injury within the 21 days prior to commencing study treatment;
* Clinically significant gastrointestinal bleeding within 6 months prior to first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-11; Primary Completion 2013-04 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Versola, Study Director — Quintiles, Inc.
Locations (19):
- United States (9):
  - Arizona Oncology Associates, PC - CASA, Tucson, Arizona
  - Boca Raton Clinical Research Associates, Inc, Plantation, Florida
  - Robert H. Lurie Comprenhensive Cancer Center of Northwestern University, Chicago, Illinois
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Medical Center, Detroit, Michigan
  - University of North Carolina at Chapel Hill, Chapell Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Mercy Cancer Centerr at St. Anne, Toledo, Ohio
- Russia (3):
  - Chelyabinsk Regional Oncology Dispensary, Chelyabinsk
  - GOU VPO St-Petersburg SMA n/a Mechnikov Fed. Agen. of Healthcare and Social Developm., Saint Petersburg
  - FSI "SRC of Oncology n. a. N.N.Petrov of Rosmedtekhnologiy", Saint Petersburg
- Ukraine (4):
  - SI Dnipropetrovsk Medical Academy of MOHU ch of Oncology and Medical Radiology, Dnipropetrovsk
  - Municipal Clinical Medical and Prophylactic Institution Donetsk Regional Antitumor Centre, Donetsk
  - Kyiv City Clinical Oncological Center, Kyiv
  - Lviv State Oncol. Reg. Treatment and Diagnostic Center, Lviv
- United Kingdom (3):
  - Barts and the London NHS Trust, London, Greater London
  - Sarah Cannon Research UK, London, Greater London
  - The Christie NHS Foundation Trust, Manchester, Greater Manchester

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were to only participate in either the Phase 1b or Phase 2 portion of the study.
Groups:
- Phase 1b: Golvatinib+Capecitabine+Cisplatin: Oral golvatinib (200 mg) was taken at about the same time each day of every 21-day treatment cycle, with or without food. Oral capecitabine (1000 mg/m^2 tablet) was taken twice a day (2000 mg/m^2 total daily) with food at about the same time (after golvatinib), on Days 1 through 14 of each 21-day cycle. At least 2 hours after capecitabine was taken, cisplatin (80 mg/m^2) was administered by intravenous (IV) infusion over 60 minutes (after appropriate hydration or according to the institutional guidelines), on Day 1 of each 21-day cycle. Pretreatment hydration included 1 liter of normal saline by IV infusion over 120 minutes. Posttreatment hydration included 500 mL normal saline over 60 minutes. The dose level of golvatinib was to be escalated (to 300 and 400 mg) for additional cohorts after 3 participants enrolled into a given cohort unless there was a dose-limiting toxicity (DLT) in the first 3 participants.
- Phase 2: Golvatinib+Capecitabine+Cisplatin: The dose of golvatinib was to be the maximum tolerated dose (MTD) as determined during the Phase 1b portion of the study in combination with capecitabine and cisplatin as described for Phase 1b.
  The study was terminated prior to Phase 2.
- Phase 2: Capecitabine + Cisplatin: Oral capecitabine (1000 mg/m^2 tablet) was taken twice a day (2000 mg/m^2 total daily) with food at about the same time (after golvatinib), on Days 1 through 14 of each 21-day cycle. At least 2 hours after capecitabine was taken, cisplatin (80 mg/m^2) was administered by intravenous (IV) infusion over 60 minutes (after appropriate hydration or according to the institutional guidelines), on Day 1 of each 21-day cycle. Pretreatment hydration included 1 liter of normal saline by IV infusion over 120 minutes. Posttreatment hydration included 500 mL normal saline over 60 minutes.
Period: Phase 1b
Arm/Group | Phase 1b: Golvatinib+Capecitabine+Cisplatin | Phase 2: Golvatinib+Capecitabine+Cisplatin | Phase 2: Capecitabine + Cisplatin
Started | 7 (Replaced 1 subject; who discontinued study drug in first cycle) | 0 | 0
Completed | 1 (The subject who completed 6 cycles was withdrawn by sponsor request.) | 0 | 0
Not Completed | 6 | 0 | 0
Not completed — Death | 4 | 0 | 0
Not completed — Study terminated by sponsor | 2 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1b: Golvatinib+Capecitabine+Cisplatin | Phase 2: Golvatinib+Capecitabine+Cisplatin | Phase 2: Capecitabine + Cisplatin
Started | 0 (Treatment arm not designated for phase 2.) | 0 (The study was terminated prior to enrollment) | 0 (The study was terminated prior to enrollment)
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Phase 1b: Golvatinib+Capecitabine+Cisplatin
Number analyzed (Participants) | 7
Age, Customized [Number; unit: Participants]
  Age range 47 to 80 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Area Under The Concentration-Time Curve (AUC) From 0 to 24 Hours of Golvatinib
Description: On days when pharmacokinetic (PK) samples were to be drawn, a predose blood sample was obtained prior to administration of golvatinib and capecitabine. After administration of study drugs, a second postdose blood sample was taken. The amount of golvatinib in the participant's blood was analyzed and the AUC was calculated. The AUC reflects the actual body exposure to drug after administration of a dose of the drug and is dependent on the rate of elimination of the drug from the body and the dose administered. Predose samples that were below the limit of quantitation (BLQ) or missing were assigned a numerical value of zero for the calculation of AUC. Any other BLQ concentrations were assigned a value of zero. Results were expressed in nanograms·hour/milliter (ng·h/mL).
Time Frame: Cycle 1 (Day -2); predose, 30 minutes, 1, 2, 3, 4, 8, 12 (if feasible), 24, and 48 hours after study treatment. Cycle 2 (Day 1); predose, 30 minutes, 1, 2, 3, 4, 8, 12 (if feasible), and 24 hours after study treatment.
Population: Pharmacokinetic (PK) population: All participants in the Safety Population who had sufficient concentration data to derive one or more of the PK parameters. Participants with partial data were evaluated on a case-by-case basis to determine if sufficient data were available for meaningful PK analysis.
Measure: Median (Full Range); unit: ng·h/mL
Arm/Group | Phase 1b: Golvatinib+Capecitabine+Cisplatin
Number analyzed (Participants) | 7
ng·h/mL
  Cycle 1, Day -2 | 23400 [5000 to 56100]
  Cycle 2, Day 1 | 26300 [17400 to 62400]

2. Primary Outcome: Maximum Concentration (Cmax) of Golvatinib
Description: Blood samples were drawn to analyze the amount of golvatinib in the participant's serum. Maximum concentration refers to the maximum (or peak) serum concentration of study drug in the participant's system after administration of the study drug and prior to the administration of a second dose of the study drug. Results were expressed in nanograms/milliliter (ng/mL).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: ng/mL
Groups:
- Phase 1b: Golvatinib+Capecitabine+Cisplatin: Oral golvatinib (200 mg) was taken at about the same time each day of every 21-day treatment cycle, with or without food. Oral capecitabine (1000 mg/m^2 tablet) was taken twice a day (2000 mg/m^2 total daily) with food at about the same time (after golvatinib), on Days 1 through 14 of each 21-day cycle. At least 2 hours after capecitabine was taken, cisplatin (80 mg/m^2) was administered by IV infusion over 60 minutes (after appropriate hydration or according to the institutional guidelines), on Day 1 of each 21-day cycle. Pretreatment hydration included 1 liter of normal saline by IV infusion over 120 minutes. Posttreatment hydration included 500 mL normal saline over 60 minutes. The dose level of golvatinib was to be escalated (to 300 and 400 mg) for additional cohorts after 3 participants enrolled into a given cohort unless there was a DLT in the first 3 participants.
Arm/Group | Phase 1b: Golvatinib+Capecitabine+Cisplatin
Number analyzed (Participants) | 7
ng/mL
  Cycle 1, Day -2 | 1680 [268 to 3890]
  Cycle 2, Day 1 | 1620 [834 to 3430]

3. Primary Outcome: Number of Participants With a Treatment-Emergent Adverse Event (TEAE)
Description: Safety assessments consisted of monitoring and recording all adverse events (AEs) and serious AEs; regular monitoring of hematology, blood chemistry, and urine values; periodic measurement of vital signs and electrocardiograms (ECGs); and performance of physical examinations. A TEAE was defined as an adverse event (AE) that had an onset date, or a worsening in severity from Baseline (pretreatment), on or after the first dose of study drug up to 30 days after the date of last study treatment.
Time Frame: From date of first dose up to 30 days after the last dose of study treatment, up to approximately 1 year 1 month.
Population: Safety Population included all participants who received at least one dose of study drug and who had at least one safety assessment after the first dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Phase 1b: Golvatinib+Capecitabine+Cisplatin
Number analyzed (Participants) | 7
Participants | 7

4. Primary Outcome: Time to Maximum Concentration (Tmax) of Golvatinib
Description: Tmax was defined as the time at which Cmax was observed for golvatinib in combination with cisplatin and capecitabine.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Phase 1b: Golvatinib+Capecitabine+Cisplatin
Number analyzed (Participants) | 7
Hours
  Cycle 1, Day -2 | 3.00 [1.00 to 7.78]
  Cycle 2, Day 1 | 6.07 [3.00 to 12.82]

5. Secondary Outcome: Overall Response Rate (ORR)
Description: The study was terminated prior to enrollment in Phase 2 so this outcome measure was not conducted.
Time Frame: Until disease progression or death for 3 years
Population: The study was terminated prior to enrollment in Phase 2 so this outcome measure was not conducted.
Groups:
- Phase 2: Capecitabine + Cisplatin: The dose of golvatinib was to be the MTD as determined during the Phase 1b portion of the study in combination with capecitabine and cisplatin as described for Phase 1b.
  The study was terminated prior to Phase 2.
Arm/Group | Phase 2: Golvatinib+Capecitabine+Cisplatin | Phase 2: Capecitabine + Cisplatin
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Time to Progression (TTP)
Description: The study was terminated prior to enrollment in Phase 2 so this outcome measure was not conducted.
Time Frame: Until disease progression or death for 3 years
Population: The study was terminated prior to enrollment in Phase 2 so this outcome measure was not conducted.
Groups:
- Phase 2: Golvatinib+Capecitabine+Cisplatin; Phase 2: Capecitabine + Cisplatin: The dose of golvatinib was to be the MTD as determined during the Phase 1b portion of the study in combination with capecitabine and cisplatin as described for Phase 1b.
  The study was terminated prior to Phase 2.
Arm/Group | Phase 2: Golvatinib+Capecitabine+Cisplatin | Phase 2: Capecitabine + Cisplatin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From date of first dose up to 30 days after the last dose of study treatment, up to approximately 1 year 1 month.
Description: Safety population included all participants enrolled in Phase 1b of this study, except for those who (a) dropped out prior to receiving study drug, or (b) were without any safety assessments after the first dose of study drug. Treatment-emergent AEs, (onset date or worsening in severity from baseline after first dose of study drug), were reported.
Arm/Group | Phase 1b: Golvatinib+Capecitabine+Cisplatin
Serious Adverse Events (participants affected / at risk) | 5/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Golvatinib+Capecitabine+Cisplatin (N=7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Psoas abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pulmonary embolism (Vascular disorders) | 1
Convulsion (Nervous system disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Golvatinib+Capecitabine+Cisplatin (N=7)
Nausea (Gastrointestinal disorders) | 7
Dehydration (Metabolism and nutrition disorders) | 5
Fatigue (General disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Decreased appetite (Metabolism and nutrition disorders) | 4
Palmar-Plantar erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 4
Anaemia (Blood and lymphatic system disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 3
Headache (Nervous system disorders) | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 3
Anxiety (Psychiatric disorders) | 2
Asthenia (General disorders) | 2
Chest pain (General disorders) | 2
Chills (General disorders) | 2
Contusion (Injury, poisoning and procedural complications) | 2
Dizziness (Metabolism and nutrition disorders) | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2
Insomnia (Psychiatric disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Pyrexia (General disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Weight decreased (Investigations) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Abdominal tenderness (Gastrointestinal disorders) | 1
Ageusia (Nervous system disorders) | 1
Amnesia (Nervous system disorders) | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Balance disorder (Nervous system disorders) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Breath sounds abnormal (Investigations) | 1
Catatonia (Psychiatric disorders) | 1
Cold sweat (General disorders) | 1
Convulsion (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Depression (Psychiatric disorders) | 1
Diaphragmatic paralysis (Respiratory, thoracic and mediastinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Electrocardiogram st segment elevation (Investigations) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Eye discharge (Eye disorders) | 1
Feeling cold (General disorders) | 1
Feeling hot (General disorders) | 1
Glossodynia (Gastrointestinal disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1
Lacrimation increased (Eye disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Malaise (General disorders) | 1
Mood swings (Psychiatric disorders) | 1
Mucosal inflammation (General disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Neuralgia (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Oedema peripheral (General disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Oropharyngeal candidiasis (Infections and infestations) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pain (General disorders) | 1
Pallor (General disorders) | 1
Palpitations (Cardiac disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Pneumonia (Infections and infestations) | 1
Proctalgia (Gastrointestinal disorders) | 1
Psoas abscess (Musculoskeletal and connective tissue disorders) | 1
Pulmonary embolism (Vascular disorders) | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Restlessness (Psychiatric disorders) | 1
Scab (Skin and subcutaneous tissue disorders) | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Streptococcal bacteraemia (Infections and infestations) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1
Trigeminal neuralgia (Nervous system disorders) | 1
Urinary tract infection (Infections and infestations) | 1
Vision blurred (Eye disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated prior to enrollment in Phase 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other